CLINICAL TRIAL: NCT04574765
Title: A Research Platform to Screen and Protect Individuals That Work Within a Food Production, Healthcare, Research or Clinical Organization - RESPECT
Brief Title: A Research Platform to Screen Healthcare Workers- Coordinated Approach to Pandemic Trials of COVID-19
Acronym: RESPECT
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: OZUHN-001; 20-5289 (Other: University Health Network)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Healthcare Worker; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Mental Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swabs Optional blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1 (A and B): Cohort 1A included health care workers. Cohort 1B includes individuals that work within a healthcare, research or clinical organization.
  Interventions: Diagnostic Test: Nasopharyngeal swab; Other: Questionnaire collection (CITF); Other: Optional blood collection; Other: Optional questionnaire completion (mental health); Diagnostic Test: Optional saliva sample (for validation); Diagnostic Test: Nasal Swab (rapid antigen test)
- Cohort 2: Cohort 2 includes Individuals that work within a food production organization.
  Interventions: Diagnostic Test: Nasopharyngeal swab; Other: Questionnaire collection (CITF); Other: Optional blood collection; Other: Optional questionnaire completion (mental health); Diagnostic Test: Optional saliva sample (for validation)
- Cohort 3: Cohort 3 includes individuals that work within a healthcare, research or clinical organization that will be tested via nasal swab only, with increased frequency of testing.
  Interventions: Diagnostic Test: Nasopharyngeal swab; Other: Optional blood collection; Other: Optional questionnaire completion (mental health); Diagnostic Test: Optional saliva sample (for validation); Diagnostic Test: Nasal Swab (rapid antigen test)

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab — Nasopharyngeal swab for COVID-19
Other: Questionnaire collection (CITF) — Fill out questionnaires regarding exposures and travel history, occupation category, any symptoms in the past 21 days, any face-to-face care of a known COVID-19 positive patients in past 14 days or any children at home who are less than 12 years of age.
  Other Names: COVID-19 Immunity Task Force (CITF)
  Groups: Cohort 1 (A and B); Cohort 2
Other: Optional blood collection — Provide blood samples to look for COVID-19 specific antibodies and/or proteins at the time of enrollment and after 8 weeks.
Other: Optional questionnaire completion (mental health) — Fill out an optional mental health questionnaire.
Diagnostic Test: Optional saliva sample (for validation) — Provide saliva sample anonymously.
Diagnostic Test: Nasal Swab (rapid antigen test) — Panbio nasal swab rapid antigen test
  Groups: Cohort 1 (A and B); Cohort 3

SUMMARY:
Recent studies have shown that some individuals may be asymptomatic but continue to shed the COVID-19 virus. These individuals may represent a population that can unknowingly transmit the virus. Healthcare workers (HCW) may acquire COVID-19 from the community or from possibly infected patients. It is important to gather data with respect to this to further understand the prevalence of asymptomatic carriage in individuals who work in research facilities, offices and clinical areas of hospitals and research facilities/institutes since this has important implications for infection control, as well as staff and patient safety. The purpose of this study is to test whether a proportion of these individuals may be asymptomatic shedders of the COVID-19 virus.

DETAILED DESCRIPTION:
Healthcare workers of participating institutions who agree to be participants will:

* Fill out some information about participants into a database portal system. Participants will have the ability to check their COVID-19 test results via the portal.
* Have nasopharyngeal (NP) swabs done for COVID-19 testing. This can be done about once a week for up to 8 weeks (about 1-8 swabs total).
* Provide optional blood samples to look for COVID-19 specific antibodies and/or proteins at the time of enrollment and after 8 weeks.
* Fill out questionnaires about participant exposures and travel history, occupation category, any symptoms in the past 21 days, whether they have provided any face-to-face care of a known COVID-19 positive patients in past 14 days or if participants have any children at home who are less than 12 years of age.
* Fill out an optional questionnaire about their mental health
* Be contacted by telephone if participants are tested positive, to determine whether participants have symptoms of COVID-19, and for the results of any follow-up COVID-19 testing that may have been done.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who work within a food production, healthcare, research or clinical organization.
* Asymptomatic as per daily screening.
* No contraindication to performing a NP swab.

Exclusion Criteria:

* Any individual with fever, respiratory or flu-like symptoms will not be eligible. Symptom positive individuals who were not picked up at entry screening will be referred to their Occupational Health. Specific symptoms include:

  * Fever, chills or headache
  * New or worsening cough
  * Shortness of breath, difficulty breathing, sore throat or difficulty swallowing
  * Runny nose or stuffy nose without another cause (e.g. allergies)
  * Nausea/vomiting, diarrhea, stomach pain
  * Decrease/loss of taste or smell
  * Unexplained fatigue, malaise, muscle aches
  * Eye pain or pink eye In addition to those symptoms listed above, individuals should also be screened for symptoms as per their institutional requirements.
* Enrolled in a COVID-related interventional study (eg. Behavioural or drug study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who work within a food production, healthcare, research or clinical organization.
Sampling Method: Non-Probability Sample
Enrollment: 7373 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Percentage of healthcare workers who are asymptomatic while COVID-19 positive | 2 years
  To determine whether asymptomatic individuals who work within a food production, healthcare, research or clinical organizationmay shed CoV during the pandemic. We hypothesize that a small proportion (~1-10%) of these asymptomatic individuals may be CoV+ either because they are in the incubation period prior to symptoms or remain asymptomatic for the duration of infection.

SECONDARY OUTCOMES:
Prevalence of any COVID-19 variants of concern in asymptomatic workers | 2 years
  To assess the prevalence of any COVID-19 variants of concern in asymptomatic workers.
Spread of any COVID-19 variants of concern in asymptomatic workers | 2 years
  To help determine the validity of the Panbio COVID-19 Ag Rapid Test and the saliva sample COVID-19 test by conducting these tests alongside the NP swab test.

CONTACTS AND LOCATIONS:
Overall Officials: Amit M Oza, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: RESEARCH ARTICLE — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0247258